CLINICAL TRIAL: NCT00158886
Title: A Phase I Study of Oral Topotecan as a Radiosensitizing Agent in Patients With Rectal Cancer
Brief Title: Oral Topotecan As A Radiosensitizing Agent In Rectal Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 104864/517
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Carcinoma, Renal Cell
Keywords: oral topotecan rectal cancer pelvic radiation
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Topotecan; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Subjects with rectal cancer (Experimental): Subjects will be administered topotecan along with concomitant radiation for five days per week for five weeks. Topotecan doses will start at 0.25 milligrams per square meter (mg/m˄2) and will be escalated 0.15 mg/m˄2 for subsequent cohorts. To advance to the next dose level of topotecan, at least two subjects will have to complete therapy with oral topotecan without experiencing grade 3 or 4 toxicity for three weeks after the oral topotecan treatment.
  Interventions: Drug: Topotecan; Radiation: Radiation therapy

INTERVENTIONS:
Drug: Topotecan — Topotecan will be provided as capsules for oral administration and will be administered at least 3 hours before radiation therapy.
  Other Names: Hycamtin
Radiation: Radiation therapy — For radiation therapy, subjects will receive 180 centigray (cGy) per fraction to a total dose of 4500 cGy to the pelvis using a 3 or 4 field technique and high energy photons (>=6 megavolt [mv]).

SUMMARY:
Patients with rectal cancer who are candidates for pre-operative radiation therapy may be enrolled in the Phase I, single center study. Patients will have a full blood count, biochemistry, urinalysis, and ECG for safety evaluation. Sequential cohorts of three patients will be given increasing doses of oral topotecan and fixed doses of concurrent radiation (45 Gy) over five weeks. The starting dose of oral topotecan is 0.25 mg/m2 to be concomitantly administered with radiation (45 Gy) x 5 days every week unless the radiation is interrupted for Holidays/Weekends or toxicity requiring treatment delays occurs. A total of 25 doses are planned.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed rectal cancer.
* Candidates for preoperative radiotherapy.
* Primary tumor at least 3cm and clinical stage of T2, T3, or T4 and any N according to the Astler-Coller modification of the Dukes staging system.
* Eastern Cooperative Oncology Group (ECOG) performance status less than 2.
* Diagnosis of rectal cancer should be no more than 90 days from start of therapy.
* Evaluation at the H. Lee Moffitt Cancer Center.
* Recovery from prior surgery and life expectancy at least 3 months.

Exclusion Criteria:

* A primary tumor totally excised.
* Recurrent rectal cancer that failed initial treatment.
* Exposure to topotecan, infection, immunodeficiencies, conditions of the gastrointestinal (GI) tract which would affect absorption, medication that maintains motility/gastric emptying.
* Any concomitant malignancy within the last five years.
* Severe medical problems unrelated to the malignancy which would limit compliance with the study.
* Patients of child bearing potential.
* Not practicing adequate contraception.
* Patients who are pregnant or lactating.
* Use of an investigational drug within 30 days or 5 half-lives of the first dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2001-11-08 (Actual); Primary Completion 2006-08-11 (Actual); Study Completion 2006-08-11 (Actual)

PRIMARY OUTCOMES:
To determine the MTD of oral topotecan in combination with pelvic radiation | Up to 24 months

SECONDARY OUTCOMES:
To evaluate the toxicity and potential efficacy of oral topotecan and concurrent pelvic radiation for the treatment of rectal cancer. To determine pathologic response to treatment and assessment of sphincter preservation. | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Tampa, Florida, United States

REFERENCES:
- See also: Results for study 104864/517 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/104864/517?search=study&search_terms=104864%2F517#rs